CLINICAL TRIAL: NCT00776789
Title: Effect of Early Skin to Skin Contact on Breast Feeding Behaviour in Term Newborns: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Anu Thukral, Doctor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: dranuthukral
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Breastfeeding
Keywords: Skin to skin contact; Salivary cortisol; Breast feeding Behavior
MeSH Terms: conditions — Breast Feeding | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- skin to skin contact (Experimental): Infants randomized to this group were placed prone over the mother's chest immediately after birth. Skin-to-skin contact was continued for the next two hours. Mothers in both the groups received support for initiating breastfeeding, if required. All mothers, regardless of the group allocation, were advised to give exclusive breastfeeding to their infants during the hospital stay. They were discouraged from giving supplemental feeds to their infants unless indicated by the duty registrar. All the mothers were counseled regarding the duration of exclusive breastfeeding at the time of discharge.
  Interventions: Other: skin to skin contact
- Control group (Experimental): The infants who were allocated to the conventional care (control group) were kept by the mother's side and did not receive early SSC. All mothers, regardless of the group allocation, were advised to give exclusive breastfeeding to their infants during the hospital stay. They were discouraged from giving supplemental feeds to their infants unless indicated by the duty registrar. All the mothers were counseled regarding the duration of exclusive breastfeeding at the time of discharge.
  Interventions: Other: Control group

INTERVENTIONS:
Other: skin to skin contact — Infants randomized to SSC group were placed prone over the mother's chest immediately after birth. Skin-to-skin contact was continued for the next two hours. breastfeeding at the time of discharge.
  Arms: skin to skin contact
Other: Control group — The infants who were allocated to the conventional care (control group) were kept by the mother's side and did not receive early SSC.
  Other Names: Conventional care
  Arms: Control group

SUMMARY:
Aims and Objectives

Aim

To determine the effect of delivery room Skin To Skin contact on breast feeding behavior of term neonates born by normal vaginal delivery at 36-48 hours.

Objectives Primary objective To determine the effect of delivery room Skin To Skin contact on breast feeding behaviour of term neonates born by normal vaginal delivery, between 36-48 hours (as measured by Infant Breast Feeding Score) by video recording using a randomized controlled design.

Secondary objectives To determine the effect of delivery room Skin to Skin contact on

1. Salivary cortisol at 6 hours as measured by electrochemiluminescence immunoassay (ECLIA)
2. Weight at 48 hours as measured by digital infant weighing scale.
3. Maternal perception of breast milk output, breast consistency, infant's feeding and activity at 36-48 hours as measured by a score graded as very satisfied, satisfied, acceptable and not satisfied.
4. Number and duration of feeding sessions till 48 hrs according to the mother as assessed at 48 hours
5. Breast feeding rates at 6 weeks measured at the time of vaccination at the time of visit to the hospital for the same or as asked by telephonic conversation.

Hypothesis

Infants receiving skin to skin contact when compared with neonates not receiving it, demonstrate better breast feeding behaviour.

DETAILED DESCRIPTION:
Inclusion and exclusion criteria for the enrollment of subjects in the study

Inclusion criteria Term babies born to mothers by normal vaginal delivery in the study period.

Exclusion criteria

1. Babies with major congenital malformation.
2. Multiple pregnancy
3. Babies requiring resuscitation beyond the initial steps
4. Babies requiring care in the neonatal intensive care unit.
5. Maternal problems requiring immediate care

   * Severe preeclampsia defined as Blood pressure more than 160/110, Proteinuria more than 3+, Oliguria less than 500 ml, Pulmonary edema, cerebral visual disturbances, Impaired liver function, Thrombocytopenia, Epigastric Pain
   * Imminent eclampsia
   * Severe bleeding
   * Mother with significant surgical or medical illness requiring separation of the baby from the mother.
6. Small for dates and large for dates babies
7. Infants of diabetic mother
8. Maternal refusal of consent

Outcome Measures:

1. Measurement of Breast feeding Behavior at 36-48 hours using Infant Breast feeding Behavior scale
2. Salivary Cortisol
3. Weight at birth
4. Weight at 48 hours
5. Number of feeding sessions till 48 hours
6. Maternal Perception of Infant activity, feeding and breast milk output.

ELIGIBILITY:
Inclusion Criteria:

* Term babies born to mothers by normal vaginal delivery in the study period.

Exclusion Criteria:

1. Babies with major congenital malformation.
2. Multiple pregnancy
3. Babies requiring resuscitation beyond the initial steps
4. Babies requiring care in the neonatal intensive care unit.
5. Maternal problems requiring immediate care

   * Severe preeclampsia defined as Blood pressure more than 160/110, Proteinuria more than 3+, Oliguria less than 500 ml, Pulmonary edema, cerebral visual disturbances, Impaired liver function, Thrombocytopenia, Epigastric Pain
   * Imminent eclampsia
   * Severe bleeding
   * Mother with significant surgical or medical illness requiring separation of the baby from the mother.
6. Small for dates and large for dates babies
7. Infants of diabetic mother
8. Maternal refusal of consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Kr Paul, MD, Study Director — All India Institute of Medical Sciences
Locations (1):
- AIIMS, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Thukral A, Sankar MJ, Agarwal R, Gupta N, Deorari AK, Paul VK. Early skin-to-skin contact and breast-feeding behavior in term neonates: a randomized controlled trial. Neonatology. 2012;102(2):114-9. doi: 10.1159/000337839. Epub 2012 Jun 14. PMID 22699241

RESULTS

PARTICIPANT FLOW:
Groups:
- Skin to Skin Contact: Babies in this arm will be given skin to skin contact for at least 2 hours after birth
- Control Group: baby will be kept by the mothers side and not given skin to skin contact
Period: Overall Study
Arm/Group | Skin to Skin Contact | Control Group
Started | 20 | 21
Completed | 17 | 18
Not Completed | 3 | 3
Not completed — Consent refusal | 2 | 2
Not completed — Poor quality video | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Skin to Skin Contact | Control Group | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 21 | 41
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] — gestation age in weeks
  weeks | 38 (0.91) | 38 (1.2) | 38 (0.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: The Median Breast Feeding Score
Description: This was a one point assessment done at 36-48 hours by video recording. The video recording was carried out in a separate well lighted room after taking informed consent from the mother. The mother had full right to see the video and only if she was satisfied, was then the video finally stored. These videos were analyzed later using the infant breast feeding assessment tool : a scoring measure [0 to 3] for i) readiness to feed ii) sucking iii) rooting and iv) latching. The total possible score could vary from 0 to 12, with 12 being the best possible total score. Successful breastfeeding was defined as a total score of more >=8.
Time Frame: 36-48 hours by video recording
Measure: Median (Inter-Quartile Range); unit: scores
Arm/Group | Skin to Skin Contact | Control Group
Number analyzed (Participants) | 17 | 18
scores | 8 [5 to 10] | 9 [5 to 10]

2. Secondary Outcome: Salivary Cortisol
Description: Saliva samples were collected with a Salivette. The infant had to suck on the swab for atleast 5 minutes. The prerequisite for collection of the saliva included that the infant should not have fed atleast 2 hours prior to the collection of the salivary sample. The filtrates were then transferred to a separate tube and were stored at 2-8º C for 24 hours. They were later transported to the central laboratory where the samples were stored at -20ºC and later analyzed using electrochemiluminescence immunoassay (ECLIA).
Time Frame: 6 hours
Measure: Median (Inter-Quartile Range); unit: microgram/dl
Arm/Group | Skin to Skin Contact | Control Group
Number analyzed (Participants) | 20 | 21
microgram/dl | 0.90 [0.35 to 2.1] | 0.54 [0.25 to 0.86]
Statistical Analysis 1: Comparison: Skin to Skin Contact vs Control Group; Test type: Superiority or Other; p = 0.4, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Breast Feeding Status at 48 Hours
Description: The mother was given a form at the time of birth of the baby for recording the duration of each breast feeding session and documentation of any supplemental feeds taken from the neonatal intensive care unit. The number and the amount of supplemental feeds was confirmed with the nursing staff on duty when in the hospital and with the mother at 6 weeks when she reported for the first vaccination or by telephonic contact with her at 6 weeks. This was recorded by the principal investigator and crosschecked by the second investigator in all cases.
Time Frame: 48 hours
Population: EBF rates were assessed using the standard WHO definitions. We asked the mothers about the method of feeding and the number and amount of supplemental feeds received in the first 2 days of life. Breastfeeding rates at 6 weeks were obtained by enquiring from the mothers at the time of the first vaccination of their infants in the follow-up clinic.
Measure: Number; unit: percentage of partcipants
Groups:
- Control Group: Babies will be kept by the mothers side and not given skin to skin contact
Arm/Group | Skin to Skin Contact | Control Group
Number analyzed (Participants) | 20 | 21
percentage of partcipants | 95 | 38
Statistical Analysis 1: Comparison: Skin to Skin Contact vs Control Group; Exclusive breast feeding at 48 hours was 95% (19 out of 20 partcipants were exclusively breast feeding)in the skin-to-skin contact group vs. 38.1% in the control group; Test type: Superiority or Other; p = 0.00, Wilcoxon (Mann-Whitney); Odds Ratio (OR) = 2.5, 95% CI [1.4 to 4.3]

4. Secondary Outcome: Breast Feeding Status at 6 Weeks
Description: as for outcome 3
Time Frame: 6 weeks
Measure: Number; unit: percentage of partcipants
Arm/Group | Skin to Skin Contact | Control Group
Number analyzed (Participants) | 20 | 21
percentage of partcipants | 90 | 28
Statistical Analysis 1: Comparison: Skin to Skin Contact vs Control Group; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney); Odds Ratio (OR) = 2.5, 95% CI [1.6 to 6.3]

ADVERSE EVENTS:
Arm/Group | Skin to Skin Contact | Control Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

LIMITATIONS AND CAVEATS:
This study evaluated breast feeding behaviour of term neonates with only one video, which may not have been an accurate marker of feeding behavior.There could a possibility of inadvertent bias at the time of intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No